CLINICAL TRIAL: NCT02526810
Title: Comparison of Glycaemic Fluctuation and Oxidative Stress Between Two Short-term Therapies for Type 2 Diabetes
Acronym: COGFOST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Guangdong Provincial Department of Science and Technology (Unknown)
Responsible Party: Principal Investigator, Longyi Zeng, Head of Endocrinology and Metabolism department, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20130319c
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: glargine; continuous subcutaneous insulin injection; blood glucose control; blood glucose fluctuation; Oxidative Stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GROUP A (Active Comparator): using continuous subcutaneous insulin injection with insulin lispro, Humalog, initiating with 0.5-0.8 IU/kg.
  Interventions: Drug: insulin lispro
- GROUP B (Experimental): using glargine combined with oral drugs: insulin glargine, Lantus( initiating with 0.2 IU/kg) with metformin hydrochloride, Glucophage 500mg bid and gliclazide modified release tablets, Diamicron modified release(MR) tablets 60mg qd.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: insulin lispro — continuous subcutaneous insulin injection( insulin lispro, Humalog) to reduce blood glucose in a certain level
  Other Names: Humalog
  Arms: GROUP A
Drug: Insulin Glargine — long-acting insulin injection with metformin hydrochloride, Glucophage and gliclazide modified release tablets, Diamicron MR to reduce blood glucose in a certain level
  Other Names: Lantus
  Arms: GROUP B

SUMMARY:
The purpose of this study is to compare the blood glucose control, glycaemic fluctuation and oxidative stress for Type 2 Diabetes between two therapies, one is glargine combined with oral drugs and the other is continuous subcutaneous insulin injection.

DETAILED DESCRIPTION:
This study was a single-center, randomized, controled and prospective trial. Type 2 diabetic patients were randomized into 2 groups (Group A and Group B). Subjects in group A would be treated by using continuous subcutaneous insulin injection with insulin lispro, while subjects in group B would be treated by using glargine with oral drugs (metformin and gliclazide modified release tablets). After achieving the target glucose levels by two different approaches in 3-5 days, maintain the target glucose level for 3-5 days. Then a Medtronic dynamic blood glucose meter would be applied to the subjects for 72 hours. The clinical data, such as demographic information, present history, past history, personal history and so on were collected in the 1st day. In the 2nd day and the last day of the trial, the blood samples of the patient were collected for the Laboratory Measurements: Cr, uric acid, aminotransferase, lipid profiles, white blood cell count, N%, fasting plasma glucose, fasting C-peptide, insulin, HbA1c and standard meal test (0.5h-postprandial and 2h-postprandial blood glucose levels, C peptide and insulin, et al. The parameters of b-cell function and glycemia fluctuation were calculated and then analyzed by spss 13.0.

ELIGIBILITY:
Inclusion Criteria:

1. investigator diagnosed type 2 diabetes( 1999 WHO diagnosis criteria).
2. diagnosed as type 2 diabetes in the first time without drug therapy, or type 2 diabetes does not accept insulin in the near 3 month and duration is shorter than 10 years
3. Fasting plasma glucose ( FPG ) ≥11.1mmol/L or glycated haemoglobin (HbA1c )≥9%.
4. agree to participate the study and sign the informed consent.

Exclusion Criteria:

1. obvious failure of heart, hepatic, kidney function.
2. severe acute or chronic complications, associated diseases. or other diseases that should not use oral hypoglycemic drug.
3. women in pregnancy or planning to get pregnancy.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
mean amplitude of glycemic excursions( MAGE) | 3-5 days after patients achieving the target glucose levels, From date of randomization, assessed up to 10 days
  a Medtronic dynamic blood glucose meter was applied to the patient for 72 hours, and MAGE is calculated according to the data.

SECONDARY OUTCOMES:
glycated hemoglobin A1c | From date of randomization until the end of study, assessed up to 15 days
  changes of HbA1c before and after the intervention
glycated albumin | From date of randomization until the end of study, assessed up to 15 days
  changes of glycated albumin before and after the intervention
fasting plasma glucose, postprandial plasma glucose (30min, 120min) | From date of randomization until the end of study, assessed up to 15 days
  changes of fasting and postprandial plasma glucose before and after the intervention
Fasting C-peptide | From date of randomization until the end of study, assessed up to 15 days
  changes of Fasting C-peptide before and after the intervention
Fasting insulin | From date of randomization until the end of study, assessed up to 15 days
  changes of Fasting insulin before and after the intervention
Homa-β | From date of randomization until the end of study, assessed up to 15 days
  changes of Homa-β before and after the intervention
insulin secretion-sensitivity index | From date of randomization until the end of study, assessed up to 15 days
  changes of insulin secretion-sensitivity index before and after the intervention
disposition index | From date of randomization until the end of study, assessed up to 15 days
  changes of disposition index before and after the intervention
standard deviation of glucose level | during three days' CGMS
  standard deviation of glucose level
area under curve (AUC) when the glucose level was higher than 7.8mmol/L | during three days' CGMS
  AUC when the glucose level was higher than 7.8mmol/L
area under curve (AUC) when the glucose level was lower than 3.9mmol/L | during three days' CGMS
  AUC when the glucose level was higher than 3.9mmol/L
thiobarbituric acid reactive substance | From date of randomization until the end of study, assessed up to 15 days
  changes of thiobarbituric acid reactive substance before and after the intervention
the level of blood 8-hydroxy-2-deoxyguanosine(8-OHdG) | From date of randomization until the end of study, assessed up to 15 days
  changes of the level of blood 8-OHdG substance before and after the intervention

OTHER OUTCOMES:
the incidence of hypoglycemia | From date of randomization until the end of study, assessed up to 15 days
  the incidence of hypoglycemia, defined as blood glucose lower than 3.9mmol/L
the incidence of severe hypoglycemia | From date of randomization until the end of study, assessed up to 15 days
  defined as hypoglycemia which need other people's help or blood glucose lower than 2.8mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Zeng Longyi, professor, Principal Investigator — Endocrinology department of the Third Affiliated Hospital of Sun Yet-san University
Locations (1):
- Endocrinology department of the Third Affiliated Hospital of Sun Yet-san University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Yang W, Lu J, Weng J, Jia W, Ji L, Xiao J, Shan Z, Liu J, Tian H, Ji Q, Zhu D, Ge J, Lin L, Chen L, Guo X, Zhao Z, Li Q, Zhou Z, Shan G, He J; China National Diabetes and Metabolic Disorders Study Group. Prevalence of diabetes among men and women in China. N Engl J Med. 2010 Mar 25;362(12):1090-101. doi: 10.1056/NEJMoa0908292. PMID 20335585
- [Background] Weng J, Li Y, Xu W, Shi L, Zhang Q, Zhu D, Hu Y, Zhou Z, Yan X, Tian H, Ran X, Luo Z, Xian J, Yan L, Li F, Zeng L, Chen Y, Yang L, Yan S, Liu J, Li M, Fu Z, Cheng H. Effect of intensive insulin therapy on beta-cell function and glycaemic control in patients with newly diagnosed type 2 diabetes: a multicentre randomised parallel-group trial. Lancet. 2008 May 24;371(9626):1753-60. doi: 10.1016/S0140-6736(08)60762-X. PMID 18502299
- [Background] Mu PW, Chen YM, Lu HY, Wen XQ, Zhang YH, Xie RY, Shu J, Wang MM, Zeng LY. Effects of a combination of oral anti-diabetes drugs with basal insulin therapy on beta-cell function and glycaemic control in patients with newly diagnosed type 2 diabetes. Diabetes Metab Res Rev. 2012 Mar;28(3):236-40. doi: 10.1002/dmrr.1292. PMID 21898754
- [Background] Zeng L, Lu H, Deng H, Mu P, Li X, Wang M. Noninferiority effects on glycemic control and beta-cell function improvement in newly diagnosed type 2 diabetes patients: basal insulin monotherapy versus continuous subcutaneous insulin infusion treatment. Diabetes Technol Ther. 2012 Jan;14(1):35-42. doi: 10.1089/dia.2011.0123. Epub 2011 Aug 30. PMID 21877913
- [Background] Brun E, Zoppini G, Zamboni C, Bonora E, Muggeo M. Glucose instability is associated with a high level of circulating p-selectin. Diabetes Care. 2001 Sep;24(9):1685. doi: 10.2337/diacare.24.9.1685. No abstract available. PMID 11522721
- [Background] Muggeo M, Zoppini G, Bonora E, Brun E, Bonadonna RC, Moghetti P, Verlato G. Fasting plasma glucose variability predicts 10-year survival of type 2 diabetic patients: the Verona Diabetes Study. Diabetes Care. 2000 Jan;23(1):45-50. doi: 10.2337/diacare.23.1.45. PMID 10857967
- [Background] Reznik Y, Cohen O, Aronson R, Conget I, Runzis S, Castaneda J, Lee SW; OpT2mise Study Group. Insulin pump treatment compared with multiple daily injections for treatment of type 2 diabetes (OpT2mise): a randomised open-label controlled trial. Lancet. 2014 Oct 4;384(9950):1265-72. doi: 10.1016/S0140-6736(14)61037-0. Epub 2014 Jul 2. PMID 24998009
- [Background] Hanson RL, Pratley RE, Bogardus C, Narayan KM, Roumain JM, Imperatore G, Fagot-Campagna A, Pettitt DJ, Bennett PH, Knowler WC. Evaluation of simple indices of insulin sensitivity and insulin secretion for use in epidemiologic studies. Am J Epidemiol. 2000 Jan 15;151(2):190-8. doi: 10.1093/oxfordjournals.aje.a010187. PMID 10645822